CLINICAL TRIAL: NCT04670653
Title: National, Multicenter, Randomized, Simple-blind, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Magnólia Nasal Gel in the Treatment of Allergic Rhinitis in Participants With Age Greater Than or Equal to 12 Years.
Brief Title: Efficacy and Safety of Magnólia Nasal Gel in the Treatment of Allergic Rhinitis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMS0619 - MAGNÓLIA
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAGNÓLIA (Experimental): Two applications in each nostril, once a day.
  Interventions: Drug: MAGNÓLIA NASAL GEL
- MOMETASONE FUROATE (Active Comparator): Two applications in each nostril, once a day.
  Interventions: Drug: MOMETASONE FUROATE

INTERVENTIONS:
Drug: MAGNÓLIA NASAL GEL — Magnólia nasal gel spray
  Arms: MAGNÓLIA
Drug: MOMETASONE FUROATE — Mometasone furoate nasal spray
  Arms: MOMETASONE FUROATE

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Magnólia nasal gel in the treatment of moderate-severe persistent or moderate-severe intermittent allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree to all trial purposes by signing and dating the informed consent forms;
* Participants of both sexes, with age greater than or equal to 12 years;
* Clinical diagnosis of moderate-severe persistent or moderate-severe intermittent allergic rhinitis, according to the ARIA classification;
* Present the general status of rhinitis as moderate or severe;
* Total nasal symptom score greater than or equal to 6 points, with congestion and one or more of the other symptoms present (itching, runny nose, and sneezing) with a score greater than or equal to 2 at the screening visit;
* Present skin sensitization test to at least one aeroallergen;

Exclusion Criteria:

* Any clinical and laboratory findings that, in the judgment of the investigator, may interfere with the safety of research participants;
* History of alcohol abuse or illicit drug use;
* Participation in a clinical trial in the year before this study;
* Pregnancy or risk of pregnancy and lactating patients;
* Known hypersensitivity to the formula components used during the clinical trial;
* Participants who present other clinical forms of rhinitis, such as, but not restricted to medicated rhinitis, vasomotor and atrophic;
* Participants dependent on decongestants (nasal or oral) or receiving allergen-specific immunotherapy;
* Participants with suggestive signs of upper airways bacterial infection;
* Participants with grade II or III septum deviation and/or presence of nasal polyps or other conditions that lead to nasal obstruction;
* Concomitant chronic or intermittent use of decongestants, antihistamines, or corticosteroids by inhalation, oral, intramuscular, or intravenous;
* Concomitant use of potent topical corticosteroids.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the reflective total nasal symptom score (rESN) averaged over the entire treatment period. | 4 weeks
  The participant will answer the nasal symptom score (together with their parents or guardians, for participants with less than 18 years old) every 12 hours, in the participant's diary. The rESN will be the average of the two measurements of the day.

SECONDARY OUTCOMES:
Incidence and severity of adverse events recorded during the study. | 6 to 10 weeks